CLINICAL TRIAL: NCT03077451
Title: A Pilot Study of Nelfinavir for the Treatment of Kaposi Sarcoma
Brief Title: Nelfinavir Mesylate in Treating Patients With Kaposi Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other); University of California, Los Angeles (Other); AIDS and Cancer Specimen Resource (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-098; NCI-2016-00071 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC 098 (Other: CTEP); AMC-098 (Other: AIDS Malignancy Consortium); 2UM1CA121947 (NIH)
Record Dates: First submitted 2016-10-19; First posted 2017-03-13 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Kaposi Sarcoma; Skin Kaposi Sarcoma
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nelfinavir mesylate) (Experimental): DOSE NELFINAVIR MESYLATE: Patients receive standard dose nelfinavir mesylate PO BID for 4 weeks in the absence of PD. Patients with PD at 4 weeks proceed to high-dose nelfinavir. At week 8, if there is SD or PR, patients advance to high-dose nelfinavir mesylate. Patients discontinue standard dose nelfinavir mesylate 4 weeks after documentation of CR.
  HIGH DOSE NELFINAVIR MESYLATE: Patients with PD continue to receive high-dose nelfinavir mesylate PO BID for 4 more weeks. If there is PD documented after 4 weeks at the high dose level, nelfinavir is discontinued. If there is SD or PR, patients continue receiving nelfinavir mesylate for 16 weeks. If there is CR, patients discontinue high-dose nelfinavir mesylate 4 weeks after documentation of CR.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nelfinavir Mesylate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nelfinavir Mesylate — Given PO
  Other Names: AG1343; Viracept

SUMMARY:
This pilot phase II trial studies how well nelfinavir mesylate works in treating patients with kaposi sarcoma. Nelfinavir mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of a therapeutic escalation strategy consisting of standard dose nelfinavir (nelfinavir mesylate), followed by high dose nelfinavir, for the treatment of Kaposi sarcoma (KS) tumor lesions. With 36 evaluable participants, the null hypothesis will be rejected if 11 or more participants respond.

SECONDARY OBJECTIVES:

I. To evaluate the safety of high dose nelfinavir among participants with KS. II. To assess the effect of nelfinavir on Kaposi sarcoma-associated herpesvirus (KSHV) lytic gene expression in tumor tissue.

III. To correlate nelfinavir and the primary active metabolite, M8, concentrations with tumor response, antiviral response, and adverse effects in participants with KS.

IV. To assess the effect of nelfinavir on KSHV copy number in saliva.

TERTIARY OBJECTIVES:

I. To assess the effect of nelfinavir on KSHV copy number in PBMC and plasma. II. To assess the effect of nelfinavir on herpes simplex virus (HSV), cytomegalovirus (CMV) and Epstein-Barr virus (EBV) copy number in saliva.

OUTLINE:

STANDARD DOSE NELFINAVIR MESYLATE: Patients receive standard dose nelfinavir mesylate orally (PO) twice daily (BID) for 4 weeks in the absence of progressive disease (PD). Patients with PD at 4 weeks proceed to high-dose nelfinavir mesylate. At week 8, if there is stable disease (SD) or partial response (PR), patients advance to high-dose nelfinavir mesylate. Patients discontinue standard dose nelfinavir mesylate 4 weeks after documentation of complete response (CR).

HIGH DOSE NELFINAVIR MESYLATE: Patients with PD continue to receive high-dose nelfinavir mesylate PO BID for 4 more weeks. If there is PD documented after 4 weeks at the high dose level, nelfinavir mesylate is discontinued. If there is SD or PR, patients continue receiving nelfinavir mesylate for 16 weeks. If there is CR, patients discontinue high-dose nelfinavir mesylate 4 weeks after documentation of CR.

After completion of study treatment, patients are followed up at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven KS involving skin (with or without visceral involvement) without need for urgent cytotoxic therapy; there should be no evidence of improvement in KS in the 4 weeks immediately prior to study enrollment
* Known human immunodeficiency virus (HIV)-1 infection status, as documented by any nationally approved, licensed HIV rapid test performed in conjunction with screening (or enzyme-linked immunosorbent assay [ELISA], test kit, and confirmed by approved test at each study site; United States (U.S.) participants only: alternatively, this documentation may include a record demonstrating that another physician has documented the participant's HIV status based on either:

  * Approved diagnostic tests, or
  * The referring physician's written record that HIV infection was documented, with supporting information on the participant's relevant medical history and/or current management of HIV infection

    * Participants enrolled outside the U.S. must have a confirmatory diagnostic test sequence as appropriate per national standards, detailed as above, performed regardless of prior documented HIV status; for HIV-negative participants, testing must be performed no more than 1 month prior to study enrollment; NOTE: the term "licensed" refers to a U.S. Food and Drug Administration (FDA)-approved kit or for sites located in countries other than the United States, a kit that has been certified or licensed by an oversight body within that country and validated internally; WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment; a reactive initial rapid test should be confirmed by either another type of rapid assay or an enzyme/chemiluminescence immunoassay (E/CIA) that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 ribonucleic acid (RNA) viral load
* Participant may be either previously untreated for KS or refractory to or intolerant of any one or more prior KS therapies
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mm^3
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin: within normal limits at each study site local laboratory
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine transaminase (ALT) (serum glutamate-pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine levels =< upper limit of institutional normal; or creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal
* HIV seropositive participants must be on antiretroviral therapy (ART) with the following criteria:

  * A complete ART regimen that does not include the study drug as one of a minimum of 3 active drugs, which may include an integrase inhibitor or efavirenz in combination with nucleoside reverse-transcriptase inhibitors (NRTIs)
  * The ART regimen must not include protease inhibitor (PIs); participants must not have received a PI-based regimen for at least 4 weeks prior to enrollment
  * Participants must either have an undetectable HIV plasma ribonucleic acid (RNA), or if plasma RNA detectable, must be on the same stable regimen for a minimum of 12 weeks prior to study enrollment
  * No minimum cluster of differentiation (CD)4 count, but maximum HIV plasma RNA of 1,000 copies/mL
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study enrollment and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study enrollment or those who have not recovered from adverse events due to agents administered more than 4 weeks prior to study enrollment
* Participants who are receiving any other investigational agents
* Participants with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nelfinavir
* Participants receiving any medications or substances that have antiviral activity against KSHV or that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A (CYP3A) or cytochrome P450, family 2, subfamily C, polypeptide 19 (2C19) are ineligible; each ART regimen must be reviewed by the PI before determining eligibility to receive nelfinavir mesylate (NFV); sensitive substrates should be avoided; of the antiretroviral drugs, only delavirdine, nevirapine, cobicistat-boosted antiretrovirals (strong CYP3A4 inhibitor), maraviroc (sensitive CYP3A4 substrate), and PIs (strong CYP3A4 inhibitor) are excluded; the following drugs are also prohibited:

Strong Inhibitors of CYP3A4:

* Antibiotics: clarithromycin, erythromycin, telithromycin, troleandomycin
* HIV: non-nucleoside reverse transcriptase inhibitors (delavirdine, nevirapine), protease inhibitors (ritonavir, indinavir, lopinavir/ritonavir, saquinavir), cobicistat-boosted antiretrovirals (e.g., elvitegravir); NOTE: Clinical trials have demonstrated that there are no clinically significant drug-drug interactions between nelfinavir and the following antiretrovirals: efavirenz (strong CYP3A4 inhibitor), etravirine (strong CYP3A4 inhibitor); therefore, these antiretrovirals will not be excluded
* Antifungals: itraconazole, ketoconazole, voriconazole, fluconazole, posaconazole
* Antidepressants: nefazodone
* Antidiuretic: conivaptan
* GI: cimetidine, aprepitant
* Hepatitis C: boceprevir, telaprevir
* Miscellaneous: seville oranges, grapefruit, or grapefruit juice and/or pomelos, star fruit, exotic citrus fruits, or grapefruit hybrids

Strong Inducers of CYP3A4:

* Glucocorticoids: cortisone (> 50 mg), hydrocortisone (> 40 mg), prednisone (> 10 mg), methylprednisolone (> 8 mg), dexamethasone (> 1.5 mg)
* Anticonvulsants: phenytoin, carbamazepine, primidone, phenobarbital and other enzyme inducing anti-convulsant drugs (EIACD)
* Antibiotics: rifampin (rifampicin), rifabutin, rifapentine
* Miscellaneous: St. John's Wort, modafinil

Strong Inhibitors of CYP2C9:

* Antifungals: fluconazole; lists including medications and substances known or with the potential to interact with the CYP3A or 2C19

Drugs with KSHV antiviral activity:

* Participants receiving any medications or substances that may interfere with KSHV replication are ineligible Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the physicians' desk reference may also provide this information; as part of the enrollment/informed consent procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product; lists include medications and substances known or with the potential to interfere with KSHV replication

  * Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
  * Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with high dose nelfinavir
  * Chronic diarrhea as defined by loose or watery stools occurring more than 3 times daily at baseline lasting more than 4 weeks or not abating on condition-appropriate therapy prior to study enrollment
  * Participant is < 2 years free of another primary malignancy; exceptions include basal cell skin cancer, stage 0-I squamous cell cancer of the skin, cervical carcinoma in situ, anal carcinoma in situ
  * Use of systemic corticosteroid therapy (except for replacement doses of glucocorticoid and/or mineralocorticoid for adrenal insufficiency); inhaled or intranasal corticosteroids for allergic or bronchospastic conditions are permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soren Gantt, Principal Investigator — AIDS Malignancy Consortium
Locations (12):
- United States (10):
  - University of Miami, Miami, Florida
  - Emory University/Grady Hospital, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Benaroya Research Institute at Virginia Mason Medical Center, Seattle, Washington
- African Cancer Institute, Stellenbosch University, Cape Town, South Africa
- Uganda Cancer Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Nelfinavir Mesylate): DOSE NELFINAVIR MESYLATE: Patients receive standard dose nelfinavir mesylate PO BID for 4 weeks in the absence of PD. Patients with PD at 4 weeks proceed to high-dose nelfinavir. At week 8, if there is SD or PR, patients advance to high-dose nelfinavir mesylate. Patients discontinue standard dose nelfinavir mesylate 4 weeks after documentation of CR.
  HIGH DOSE NELFINAVIR MESYLATE: Patients with PD continue to receive high-dose nelfinavir mesylate PO BID for 4 more weeks. If there is PD documented after 4 weeks at the high dose level, nelfinavir is discontinued. If there is SD or PR, patients continue receiving nelfinavir mesylate for 16 weeks. If there is CR, patients discontinue high-dose nelfinavir mesylate 4 weeks after documentation of CR.
  Laboratory Biomarker Analysis: Correlative studies
  Nelfinavir Mesylate: Given PO
Period: Overall Study
Arm/Group | Treatment (Nelfinavir Mesylate)
Started | 36
Completed | 20
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nelfinavir Mesylate)
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 52 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 21
  More than one race | 0
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 15
  Non-Hispanic Black | 11
  Hispanic | 8
  Unknown | 2
HIV status [Count of Participants; unit: Participants]
  HIV positive | 30
  HIV negative | 6

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Therapeutic Escalation of Standard Dose Nelfinavir, Followed by High Dose Nelfinavir, for Treatment of Kaposi Sarcoma Lesions for HIV Positive Participants
Description: The binomial proportion and its exact 95% confidence interval will be used to estimate the overall response rate in the study. Overall response is defined as Complete response or partial response. Response and progression will be evaluated in this study using the AIDS Clinical Trials Groups (ACTG) response criteria for Kaposi sarcoma.
  Complete response (CR) is defined as the absence of any detectable residual disease, including tumor-associated edema, persisting for at least 4 weeks. Partial response (PR) is defined as no new lesions (skin or oral), or new visceral sites of involvement (or the appearance or worsening of tumor-associated edema or effusions); 50% or greater decrease in the number of all previously existing lesions lasting for at least 4 weeks; OR Complete flattening of at least 50% of all previously raised lesions; OR 50% decrease in the sum of the products of the largest perpendicular diameters of the marker lesions.
Time Frame: Baseline up to 16 weeks
Population: Among 30 HIV-positive patients, there are 25 HIV-positive who were treated with high dose.
Measure: Number (95% Confidence Interval); unit: percentage of overall response patients
Arm/Group | Treatment (Nelfinavir Mesylate)
Number analyzed (Participants) | 25
percentage of overall response patients | 32 [14.9 to 53.5]

2. Primary Outcome: Efficacy of Therapeutic Escalation of Standard Dose Nelfinavir, Followed by High Dose Nelfinavir, for Treatment of Kaposi Sarcoma Lesions for HIV Negative Participants
Description: The binomial proportion and its exact 95% confidence interval will be used to estimate the response rate in the study. Response rate will be estimated using the binomial proportion and it's exact 95% confidence interval for HIV negative participants.
Time Frame: Baseline up to 16 weeks
Population: There are 6 HIV-negative who were treated with high dose.
Measure: Number (95% Confidence Interval); unit: percentage of overall response patients
Arm/Group | Treatment (Nelfinavir Mesylate)
Number analyzed (Participants) | 6
percentage of overall response patients | 16.7 [0.4 to 64.1]

3. Secondary Outcome: Frequency and Severity of Adverse Events in HIV-positive Participants as Assessed by CTCAE v4.0
Description: Frequency of adverse events and their severity will be tabulated to evaluate tolerance of high dose nelfinavir in the treatment of KS in participant who are HIV-positive
Time Frame: Baseline to up to 16 weeks
Population: High dose of nelfinavir after standard dose of nelfinavir in the treatment of KS in participant who are HIV-positive. Overall Number of Participants Analyzed signifies all participants received high does of nelfinavir assessed for adverse events. Number Analyzed represents the number of participants affected with the total number of observed adverse events reported.
Measure: Number; unit: Number of adverse events
Groups:
- High Dose of Nelfinavir in the Treatment of KS in Participant Who Are HIV-positive: High dose of nelfinavir after standard dose of nelfinavir in the treatment of KS in participant who are HIV-positive
Arm/Group | High Dose of Nelfinavir in the Treatment of KS in Participant Who Are HIV-positive
Number analyzed (Participants) | 25
Number of adverse events
  Anemia: number analyzed (Participants) | 5
  Anemia | 7
  Blood and Lymphatic System Disorder: number analyzed (Participants) | 2
  Blood and Lymphatic System Disorder | 2
  Abdominal Pain: number analyzed (Participants) | 3
  Abdominal Pain | 3
  Constipation: number analyzed (Participants) | 2
  Constipation | 2
  Diarrhea: number analyzed (Participants) | 19
  Diarrhea | 42
  Nausea: number analyzed (Participants) | 7
  Nausea | 7
  Vomiting: number analyzed (Participants) | 2
  Vomiting | 2
  Edema Limbs: number analyzed (Participants) | 3
  Edema Limbs | 6
  Fever: number analyzed (Participants) | 3
  Fever | 3
  General Disorders and Administration Site Conditions: number analyzed (Participants) | 4
  General Disorders and Administration Site Conditions | 7
  Pain: number analyzed (Participants) | 4
  Pain | 6
  Herpes Simplex reactivation: number analyzed (Participants) | 2
  Herpes Simplex reactivation | 3
  Infections and Infestations: number analyzed (Participants) | 4
  Infections and Infestations | 6
  Injury, Poisoning and Procedural Complications: number analyzed (Participants) | 3
  Injury, Poisoning and Procedural Complications | 4
  Neutrophil Count Decreased: number analyzed (Participants) | 3
  Neutrophil Count Decreased | 5
  White Blood Cell Decreased: number analyzed (Participants) | 3
  White Blood Cell Decreased | 3
  Anorexia: number analyzed (Participants) | 2
  Anorexia | 2
  Hyperglycemia: number analyzed (Participants) | 3
  Hyperglycemia | 3
  Hypertriglyceridemia: number analyzed (Participants) | 4
  Hypertriglyceridemia | 5
  Arthralgia: number analyzed (Participants) | 2
  Arthralgia | 2
  Back Pain: number analyzed (Participants) | 2
  Back Pain | 2
  Musculoskeletal and Connective Tissue DIsorder: number analyzed (Participants) | 2
  Musculoskeletal and Connective Tissue DIsorder | 2
  Myalgia: number analyzed (Participants) | 2
  Myalgia | 2
  Pain in Extremity: number analyzed (Participants) | 4
  Pain in Extremity | 5
  Tumor Pain: number analyzed (Participants) | 2
  Tumor Pain | 2
  Dizziness: number analyzed (Participants) | 2
  Dizziness | 2
  Headache: number analyzed (Participants) | 2
  Headache | 2
  Insomnia: number analyzed (Participants) | 2
  Insomnia | 2
  Cough: number analyzed (Participants) | 4
  Cough | 6
  Nasal Congestion: number analyzed (Participants) | 3
  Nasal Congestion | 3
  Respiratory, Thoracic and Medastinal Disorders: number analyzed (Participants) | 3
  Respiratory, Thoracic and Medastinal Disorders | 3
  Sore Throat: number analyzed (Participants) | 4
  Sore Throat | 4
  Dry Skin: number analyzed (Participants) | 2
  Dry Skin | 2
  Pruritus: number analyzed (Participants) | 3
  Pruritus | 3
  Rash Maculo-papular: number analyzed (Participants) | 2
  Rash Maculo-papular | 2
  Skin and Subcutaneous Tissue Disorders: number analyzed (Participants) | 3
  Skin and Subcutaneous Tissue Disorders | 4
  Hypertension: number analyzed (Participants) | 5
  Hypertension | 13

4. Secondary Outcome: Frequency and Severity of Adverse Events in HIV-negative Participants as Assessed by CTCAE v4.0
Description: Frequency of adverse events and their severity will be tabulated to evaluate tolerance of high dose nelfinavir in the treatment of KS in participant who are HIV-negative
Time Frame: Baseline to up to 16 weeks
Population: High dose of Nelfinavir after standard dose among HIV-negative participants. Overall Number of Participants Analyzed signifies all participants received high does of nelfinavir assessed for adverse events. Number Analyzed represents the number of participants affected with the total number of observed adverse events reported.
Measure: Number; unit: Number of adverse events
Groups:
- High Dose of Nelfinavir in the Treatment of KS in Participant Who Are HIV-negative: High dose of nelfinavir after standard dose of nelfinavir in the treatment of KS in participant who are HIV-negative
Arm/Group | High Dose of Nelfinavir in the Treatment of KS in Participant Who Are HIV-negative
Number analyzed (Participants) | 6
Number of adverse events
  Anemia: number analyzed (Participants) | 1
  Anemia | 1
  Diarrhea: number analyzed (Participants) | 5
  Diarrhea | 9
  Flatulence: number analyzed (Participants) | 1
  Flatulence | 1
  Nausea: number analyzed (Participants) | 1
  Nausea | 1
  Chills: number analyzed (Participants) | 1
  Chills | 1
  Fatigue: number analyzed (Participants) | 1
  Fatigue | 1
  Localized Edema: number analyzed (Participants) | 1
  Localized Edema | 1
  Malaise: number analyzed (Participants) | 1
  Malaise | 1
  Fall: number analyzed (Participants) | 1
  Fall | 1
  Alanine Amino Transferase Increased: number analyzed (Participants) | 1
  Alanine Amino Transferase Increased | 1
  Aspartate Amino Transferase Increased: number analyzed (Participants) | 2
  Aspartate Amino Transferase Increased | 2
  Blood Bilirubin Increased: number analyzed (Participants) | 1
  Blood Bilirubin Increased | 1
  Creatinine Increased: number analyzed (Participants) | 1
  Creatinine Increased | 1
  Investigations: number analyzed (Participants) | 2
  Investigations | 6
  Anorexia: number analyzed (Participants) | 1
  Anorexia | 1
  Hyperglycemia: number analyzed (Participants) | 1
  Hyperglycemia | 1
  Hyperkalemia: number analyzed (Participants) | 1
  Hyperkalemia | 1
  Hypertriglyceridemia: number analyzed (Participants) | 3
  Hypertriglyceridemia | 3
  Hypoalbuminemia: number analyzed (Participants) | 1
  Hypoalbuminemia | 1
  Hypocalcemia: number analyzed (Participants) | 1
  Hypocalcemia | 1
  Hypoglycemia: number analyzed (Participants) | 1
  Hypoglycemia | 1
  Hypokalemia: number analyzed (Participants) | 1
  Hypokalemia | 5
  Hyponatremia: number analyzed (Participants) | 1
  Hyponatremia | 1
  Hypophosphatemia: number analyzed (Participants) | 1
  Hypophosphatemia | 1
  Generalized Muscle Weakness: number analyzed (Participants) | 1
  Generalized Muscle Weakness | 1
  Dizziness: number analyzed (Participants) | 2
  Dizziness | 2
  Headache: number analyzed (Participants) | 2
  Headache | 2
  Memory Impairment: number analyzed (Participants) | 1
  Memory Impairment | 1
  Insomnia: number analyzed (Participants) | 1
  Insomnia | 1
  Cough: number analyzed (Participants) | 1
  Cough | 1
  Dyspnea: number analyzed (Participants) | 1
  Dyspnea | 1
  Sore Throat: number analyzed (Participants) | 1
  Sore Throat | 1
  Hyperhidrosis: number analyzed (Participants) | 1
  Hyperhidrosis | 1
  Skin and Subcutaneous Tissue Disorders: number analyzed (Participants) | 1
  Skin and Subcutaneous Tissue Disorders | 3
  Hypertension: number analyzed (Participants) | 1
  Hypertension | 1

5. Secondary Outcome: Assess the Effect of Nelfinavir on KSHV Gene Expression in Tumor Tissue
Description: Descriptive statistics will be used for changes in the relative abundance of all latent and lytic viral mRNA relative to cellular mRNA by expression array, and changes in the percentage of cells staining for K8.1 (lytic) and LANA (latent) antigens by immunohistochemistry. Generalized estimating equations will be used to evaluate these changes over time. Normalizing transformations will be used as needed.
Time Frame: Baseline to up to 16 weeks
Population: LANA and K8.1 were reported using percentage of cells with median and IQR.
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Treatment (Nelfinavir Mesylate)
Number analyzed (Participants) | 36
percentage of cells
  LANA at baseline: number analyzed (Participants) | 13
  LANA at baseline | 10 [3 to 20]
  LANA at Day 70: number analyzed (Participants) | 6
  LANA at Day 70 | 7.5 [5 to 20]
  LANA (change): number analyzed (Participants) | 6
  LANA (change) | 0 [-5 to 0]
  K8.1 at baseline: number analyzed (Participants) | 3
  K8.1 at baseline | 3 [1 to 5]

6. Secondary Outcome: Correlate Nelfinavir and the Primary Active Metabolite, M8, Concentrations With Tumor Response, Antiviral Response, and Adverse Effects in Participants With KS.
Description: Trough nelfinavir/M8 concentrations will be summarized using descriptive statistics and 95% confidence intervals. This outcome will also be displayed graphically as a trend in drug levels over time. The relationship between dose and drug exposure of nelfinavir/M8 and the pharmacodynamic (PD) effects will be determined using Pearson's correlation coefficient (r2) or appropriate non-parametric statistics for dichotomous and categorical variables (e.g., Mann-Whitney U-test or Kruskal-Wallis analysis of variance by ranks).
Time Frame: Baseline to up to 16 weeks
Population: Participants who received study treatment. Area under the curve (AUC) of M8 measurements was reported by tumor response and adverse event grade using median and inter-quartile range (IQR).
Measure: Median (Inter-Quartile Range); unit: ng*cycle/mL
Groups:
- High Dose Treatment After Receiving the Standard Dose (Nelfinavir Mesylate): This study is not parallel arm study. Nelfinavir dose will be administrated in the sequential manner according to the response.
  AE summary is based on participants who received high dose. There were totally 31 participants received high dose after receiving standard dose.
  All patients will received standard dose of nelfinavir (1250 mg BID) for at least 4 weeks. If after 4 weeks there is progressive disease (PD), the participant will advance to the high dose nelfinavir (3125 mg BID). If by 8 weeks there is stable disease (SD) or partial response (PR) at the standard dose, the participant will advance to high dose of nelfinavir.
  The high dose nelfinavir treatment will be continued for at least 4 weeks. If there is progressive disease (PD) documented after 4 weeks at the high dose level, nelfinavir will be discontinued. If there is stable disease (SD) or partial response (PR) at the high dose level, high dose nelfinavir will be continued for up to 16 weeks. If there is a complete response (CR), high dose treatment will be discontinued 4 weeks after documentation of complete response.
- Standard Dose Treatment (Nelfinavir Mesylate): This study is not parallel arm study. Nelfinavir dose will be administrated in the sequential manner according to the response.
  AE summary is based on participants who received standard dose. There were totally 36 participants received standard dose initally.
  All patients will received standard dose of nelfinavir (1250 mg BID) for at least 4 weeks. If there is complete response (CR) at any time at the standard dose, nelfinavir will be discontinued 4 weeks after documentation of CR.
Arm/Group | High Dose Treatment After Receiving the Standard Dose (Nelfinavir Mesylate) | Standard Dose Treatment (Nelfinavir Mesylate)
Number analyzed (Participants) | 31 | 5
ng*cycle/mL
  Responders among HIV positive: number analyzed (Participants) | 9 | 0
  Responders among HIV positive | 52000 [23252 to 70075] |
  Responder among HIV negative: number analyzed (Participants) | 0 | 0
  Non-responder among HIV positive: number analyzed (Participants) | 18 | 5
  Non-responder among HIV positive | 28202 [8726 to 35372] | 0 [0 to 2513]
  Non-responder among HIV negative: number analyzed (Participants) | 4 | 0
  Non-responder among HIV negative | 80706 [6084 to 160927] |
  AE maximum grade 3+ among HIV positive: number analyzed (Participants) | 9 | 0
  AE maximum grade 3+ among HIV positive | 31402 [19605 to 69630] |
  AE maximum grade 3+ among HIV negative: number analyzed (Participants) | 2 | 0
  AE maximum grade 3+ among HIV negative | 80058 [42586 to 1175314] |
  AE maximum grade 1/2 among HIV positive: number analyzed (Participants) | 15 | 5
  AE maximum grade 1/2 among HIV positive | 30280 [11151 to 45568] | 0 [0 to 2513]
  AE maximum grade 1/2 among HIV negative: number analyzed (Participants) | 2 | 0
  AE maximum grade 1/2 among HIV negative | 92552 [49480 to 135624] |

7. Secondary Outcome: Assess the Effect of Nelfinavir on KSHV Copy Number in Saliva
Description: Pre-treatment oral samples and oral samples during treatment will be collected from each participant. The sampling frequency is irrelevant as long as the quantity is sufficient. With 36 participants, a decrease in the proportion of participants with detectable KSHV DNA from 50% at baseline to 1% on treatment can be detected at the one-sided 0.05 significance level with 0.99 power using McNemar's test.
Time Frame: Up to 16 weeks
Population: Participants who received study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nelfinavir Mesylate)
Number analyzed (Participants) | 36
Participants
  Positive swab result | 14
  Negative swab result | 20
  Unavailable swab result | 2

ADVERSE EVENTS:
Time Frame: 8 weeks (4 weeks for standard dose and 4 weeks for high dose);
Description: Among 36 participants, 31 participants received the high dose of nelfinavir after receiving the standard dose of nelfinavir.
  Mortality report was based on all 36 participants. For mortality report in high dose was based on 31 participants which is a subset of 36 participants.
  Adverse Event and Serious Adverse Event reports were based on 36 participants treated with standard dose levels of nelfinavir and 31 participants treated with high dose after standard dose.
Arm/Group | High Dose Treatment After Receiving the Standard Dose (Nelfinavir Mesylate) | Standard Dose Treatment (Nelfinavir Mesylate)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/36
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/36
Other Adverse Events (participants affected / at risk) | 28/31 | 5/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Treatment After Receiving the Standard Dose (Nelfinavir Mesylate) (N=31) | Standard Dose Treatment (Nelfinavir Mesylate) (N=36)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Treatment After Receiving the Standard Dose (Nelfinavir Mesylate) (N=31) | Standard Dose Treatment (Nelfinavir Mesylate) (N=36)
Anemia (Blood and lymphatic system disorders) | 6 (8) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 24 (51) | 3 (4)
DIZZINESS (Nervous system disorders) | 4 (4) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 2 (3) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 2 (2) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 7 (8) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 8 (8) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 4 (7) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2)
HYPERTENSION (Vascular disorders) | 6 (14) | 0 (0)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 0 (0)
EDEMA LIMBS (General disorders) | 3 (6) | 0 (0)
FEVER (General disorders) | 3 (3) | 0 (0)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 4 (7) | 0 (0)
LOCALIZED EDEMA (General disorders) | 2 (3) | 0 (0)
MALAISE (General disorders) | 2 (2) | 0 (0)
PAIN (General disorders) | 4 (6) | 0 (0)
HERPES SIMPLEX REACTIVATION (Infections and infestations) | 2 (3) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 4 (6) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER, SPECIFY (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (2) | 0 (0)
CREATININE INCREASED (Investigations) | 2 (2) | 0 (0)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 3 (7) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (5) | 0 (0)
WHITE BLOOD CELL DECREASED (Investigations) | 3 (3) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (4) | 0 (0)
INSOMNIA (Psychiatric disorders) | 3 (3) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/51/NCT03077451/Prot_SAP_ICF_000.pdf